CLINICAL TRIAL: NCT01996813
Title: The Effect of Compression Stockings on Cerebral Desaturation Events in Obese Patients Undergoing Shoulder Arthroscopy in the Beach Chair Position
Brief Title: Compression Stocking Use in Shoulder Arthroscopy in Beach Chair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Doug Evans, MD, Loyola University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 205159
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Shoulder Impingement
Keywords: arthroscopy; shoulder; obesity; beach chair; compression hose
MeSH Terms: conditions — Obesity; Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prospective Case (Experimental): Patients with a BMI of 30 kg/m^2 or greater who underwent shoulder arthroscopy in the beach chair position and were monitored intraoperatively using near-infrared spectroscopy while wearing thigh-high compression stockings.
  Interventions: Device: Thigh-high compression stockings
- Historical Control (No Intervention): Patients with a BMI of 30 kg/m^2 or greater who underwent elective shoulder arthroscopy in the beach-chair position and were monitored intraoperatively using near-infrared spectroscopy but without wearing compression stockings.

INTERVENTIONS:
Device: Thigh-high compression stockings — The intervention in this study are thigh-high compression stockings manufactured by Covidien.
  Other Names: Thrombo-Embolic Deterrent (TED) Anti-Embolism Stockings
  Arms: Prospective Case

SUMMARY:
Shoulder arthroscopy is one of the most commonly performed orthopaedic procedures and it is often done with the patient in the upright, or beach chair position (BCP). There have been multiple reported complications associated with the BCP, including cerebral ischemia, loss of vision, ophthalmoplegia, stroke, and even death. It has been reported that patients with a body mass index (BMI) of 34 or greater are as much as 12 times more likely to experience cerebral desaturation events (CDEs) compared to non-obese controls. CDEs in the upright position are hypothesized to be partially related to reduced cardiac preload due to venous pooling in the lower extremities which is exaggerated in obese patients. This prospective observational study aims to determine if the use of compression stockings in obese patients undergoing shoulder arthroscopy in the BCP can reduce the incidence, frequency, or magnitude of CDEs experienced by the patient

DETAILED DESCRIPTION:
There have been numerous studies recently in the orthopaedic surgery and anesthesia literature related to both complications associated with arthroscopy in the BCP and ongoing efforts to improve patient safety. Advantages of this position when compared with the lateral decubitus position include easier anatomic orientation, lack of traction on the brachial plexus, ease of exam under anesthesia, and easier conversion to an open approach if needed. While extremely uncommon, complications such as ischemic brain and spinal cord injury as well as visual loss and ophthalmoplegia have been reported. A recent study reported that obesity increases the likelihood of having a CDE by as many as 12 times. CDEs were defined as intra-operative decreases in regional cerebral tissue oxygen saturation (rSO2) of 20% or greater from baseline as measured by near-infrared spectroscopy (NIRS). Since obesity is so common, it was decided to investigate a measure to potentially help decrease CDEs in this population.

The exact etiology of CDEs has not been definitively demonstrated and it is felt to be multifactorial. The sympathetic nervous system normally increases systemic vascular resistance and heart rate to maintain mean arterial blood pressure (MAP) when a person sits up or stands upright. This response is blunted by the vasodilatory effects of intravenous and inhaled anesthetics used in patients undergoing shoulder arthroscopy in the BCP. The result is decreased MAP and cerebral perfusion pressure that can contribute to hypoxic brain injury. The use of sequential compression devices placed on the legs of patients undergoing shoulder arthroscopy in the BCP has been shown to reduce the incidence of hypotension by increasing cardiac preload. This study excluded obese patients (BMI > 30) and did not directly monitor rSO2, but rather only monitored hemodynamic variables.

Compression stockings are often used in patients with venous insufficiency to help with pain and to control edema. The stockings compress the soft tissues and veins, and in conjunction with sequential compression devices (SCDs), may help to increase preload in an anesthetized patient in the BCP. To our knowledge, the effect of compression stockings on cerebral perfusion has not been studied. This study aims to determine if the use of compression stockings in obese patients undergoing shoulder arthroscopy in the BCP can decrease the incidence, frequency or magnitude of CDEs as measured by NIRS. We hypothesize that the use of compression stockings will result in decreased incidence and frequency of CDEs in our population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* BMI greater than or equal to 30 kg/m^2
* Capable of receiving an interscalene nerve block.

Exclusion Criteria:

* Age < 18
* History of carotid artery stenosis equal to or greater than 90%
* History of stroke
* History of transient ischemic attack
* History of syncope
* History of vision loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2015-07-27 (Actual); Study Completion 2015-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Evans, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS, Vaughn J, Nisman M. Cerebral oxygen desaturation events assessed by near-infrared spectroscopy during shoulder arthroscopy in the beach chair and lateral decubitus positions. Anesth Analg. 2010 Aug;111(2):496-505. doi: 10.1213/ANE.0b013e3181e33bd9. Epub 2010 May 27. PMID 20508134
- [Background] Pohl A, Cullen DJ. Cerebral ischemia during shoulder surgery in the upright position: a case series. J Clin Anesth. 2005 Sep;17(6):463-9. doi: 10.1016/j.jclinane.2004.09.012. PMID 16171668
- [Background] Bhatti MT, Enneking FK. Visual loss and ophthalmoplegia after shoulder surgery. Anesth Analg. 2003 Mar;96(3):899-902. doi: 10.1213/01.ANE.0000047272.31849.F9. PMID 12598282
- [Background] Papadonikolakis A, Wiesler ER, Olympio MA, Poehling GG. Avoiding catastrophic complications of stroke and death related to shoulder surgery in the sitting position. Arthroscopy. 2008 Apr;24(4):481-2. doi: 10.1016/j.arthro.2008.02.005. PMID 18375282
- [Background] Fischer GW, Torrillo TM, Weiner MM, Rosenblatt MA. The use of cerebral oximetry as a monitor of the adequacy of cerebral perfusion in a patient undergoing shoulder surgery in the beach chair position. Pain Pract. 2009 Jul-Aug;9(4):304-7. doi: 10.1111/j.1533-2500.2009.00282.x. Epub 2009 Mar 17. PMID 19490464
- [Background] Peruto CM, Ciccotti MG, Cohen SB. Shoulder arthroscopy positioning: lateral decubitus versus beach chair. Arthroscopy. 2009 Aug;25(8):891-6. doi: 10.1016/j.arthro.2008.10.003. Epub 2008 Nov 28. PMID 19664509
- [Background] Salazar D, Sears BW, Aghdasi B, Only A, Francois A, Tonino P, Marra G. Cerebral desaturation events during shoulder arthroscopy in the beach chair position: patient risk factors and neurocognitive effects. J Shoulder Elbow Surg. 2013 Sep;22(9):1228-35. doi: 10.1016/j.jse.2012.12.036. Epub 2013 Feb 15. PMID 23415820
- [Background] Smith JJ, Porth CM, Erickson M. Hemodynamic response to the upright posture. J Clin Pharmacol. 1994 May;34(5):375-86. doi: 10.1002/j.1552-4604.1994.tb04977.x. PMID 8089249
- [Background] Kwak HJ, Lee JS, Lee DC, Kim HS, Kim JY. The effect of a sequential compression device on hemodynamics in arthroscopic shoulder surgery using beach-chair position. Arthroscopy. 2010 Jun;26(6):729-33. doi: 10.1016/j.arthro.2009.10.001. Epub 2010 Mar 3. PMID 20511029
- [Background] Hamdan A. Management of varicose veins and venous insufficiency. JAMA. 2012 Dec 26;308(24):2612-21. doi: 10.1001/jama.2012.111352. PMID 23268520
- [Background] Pollard V, Prough DS, DeMelo AE, Deyo DJ, Uchida T, Stoddart HF. Validation in volunteers of a near-infrared spectroscope for monitoring brain oxygenation in vivo. Anesth Analg. 1996 Feb;82(2):269-77. doi: 10.1097/00000539-199602000-00010. PMID 8561326
- [Derived] Tauchen AJ, Salazar D, Barton GJ, Francois A, Tonino P, Garbis NG, Evans D. The Effect of Compression Stockings on Cerebral Desaturation Events in Obese Patients Undergoing Shoulder Arthroscopy in the Beach-Chair Position. Arthroscopy. 2015 Dec;31(12):2352-64. doi: 10.1016/j.arthro.2015.06.017. Epub 2015 Aug 3. PMID 26248495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the prospective case cohort, 23 participants were recruited from December 2013 through May 2014 (6 months) from a tertiary care practice. The remaining 24 participants were historical control participants
Period: Overall Study
Arm/Group | Prospective Case | Historical Control
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises the 23 prospective cases who met inclusion criteria and were not excluded by the principal investigator as well as 24 historical control participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Historical Control | Prospective Case | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.33 (11.53) | 52.96 (10.82) | 53.15 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 16 | 11 | 27
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 47
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 35.00 [32.55 to 37.90] | 33.40 [31.20 to 36.10] | 34.30 [31.30 to 37.60]
Comorbid Diabetes [Count of Participants; unit: Participants]
  No | 19 | 19 | 38
  Yes | 5 | 4 | 9
Comorbid Peripheral Vascular Disease [Count of Participants; unit: Participants]
  No | 24 | 22 | 46
  Yes | 0 | 1 | 1
Comorbid Hypertension [Count of Participants; unit: Participants]
  No | 10 | 10 | 20
  Yes | 14 | 13 | 27
Comorbid Obstructive Sleep Apnea [Count of Participants; unit: Participants]
  No | 16 | 17 | 33
  Yes | 8 | 6 | 14
Comorbid Coronary Artery Disease [Count of Participants; unit: Participants]
  No | 21 | 22 | 43
  Yes | 3 | 1 | 4
Comorbid Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants]
  No | 22 | 22 | 44
  Yes | 2 | 1 | 3
Smoker [Count of Participants; unit: Participants]
  No | 15 | 21 | 36
  Yes | 9 | 2 | 11
Technique used to secure the airway [Count of Participants; unit: Participants]
  Endotracheal Tube | 3 | 6 | 9
  Laryngeal Mask Airway | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Desaturation Event
Description: The prevalence of a cerebral desaturation event is compared between prospective patients who underwent shoulder arthroscopy in the beach chair position while wearing thigh-high compression stockings versus historical control patients who underwent shoulder arthroscopy in the beach chair position and did not wear thigh-high compression stockings.
Time Frame: Assessed intraoperatively, an average of 114 minutes
Population: The analysis population comprises the 23 prospective cases who met inclusion criteria and were not excluded by the principal investigator as well as 24 historical control participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control | Prospective Case
Number analyzed (Participants) | 24 | 23
Participants
  No Cerebral Desaturation Event | 17 | 22
  Cerebral desaturation event | 7 | 1
Statistical Analysis 1: Comparison: Historical Control vs Prospective Case; The null hypothesis is that there is no difference in the odds of a cerebral desaturation event between patients wearing versus not wearing thigh-high compression stockings during shoulder arthroscopy in the beach chair position; Test type: Superiority; p = .0553, Regression, Logistic — The exact p-value was estimated; The method was exact logistic regression; Odds Ratio (OR) = 0.115, 95% CI 2-sided [0.002 to 1.034]

2. Secondary Outcome: Operation Time
Description: The length of operation time (in minutes) is compared between prospective patients who underwent shoulder arthroscopy in the beach chair position while wearing thigh-high compression stockings versus historical control patients who underwent shoulder arthroscopy in the beach chair position and did not wear thigh-high compression stockings.
Time Frame: End of surgery
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: Minutes
Arm/Group | Historical Control | Prospective Case
Number analyzed (Participants) | 24 | 23
Minutes | 94.08 (15.47) | 134.40 (44.44)
Statistical Analysis 1: Comparison: Historical Control vs Prospective Case; The null hypothesis is that there is no difference in the average length of surgery between patients wearing versus not wearing thigh-high compression stockings during shoulder arthroscopy in the beach chair position; Test type: Superiority; p < .001, t-test, 2 sided; A Satterthwaite correction was used to adjust the degrees of freedom; Mean Difference (Final Values) = 40.31, 95% CI 2-sided [20.22 to 60.39]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from December 2013 through May 2014 (6 months)
Description: In the historical control group, there are no participants at-risk for adverse events or all-cause mortality because they were a retrospective sample that did not receive compression stockings.
Arm/Group | Historical Control | Prospective Case
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/23

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes